CLINICAL TRIAL: NCT01843400
Title: Drug Use Investigation of Regorafenib/ STIVARGA for Unresectable, Metastatic or Recurrent Colorectal Cancer
Brief Title: Regorafenib Post-marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16472; STIVARGA-CRC-01 (Other: company internal)
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Neoplasms
Keywords: Regorafenib; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — Patients treated with Regorafenib under practical manner for colorectal cancer.

SUMMARY:
This study is a regulatory post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Regorafenib for colorectal cancer.

The objective of this study is to assess safety and effectiveness of Regorafenib using in real clinical practice.

A total of 1,250 patients are to be enrolled and assessed in 6 months standard observational period. At 12 months after the first administration of Regorafenib for confirmation of efficacy information including treatment duration and survival status of the patient.

ELIGIBILITY:
Inclusion Criteria:Patients

* who are determined to start Regorafenib/ STIVARGA treatment

Exclusion Criteria:

* Patients who have previously received Regorafenib/ STIVARGA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with unresectable, metastatic or recurrent colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 1301 (Actual)
Dates: Start 2013-04-22 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse drug reactions (ADRs) from the first administration of regorafenib | Up to 6 months
Number of patients with serious adverse events(SAEs) from the first administration of regorafenib. | up to 6 months

SECONDARY OUTCOMES:
Number of pateints with ADRs in subpopulations | Up to 6 months
Number of patients with SAEs in supopulations | Up to 6 months
Overall survival (OS) | Up to 12 months
Overall survival in subpopulations | Up to 12 months
Time to treatment failure (TTF) | Up to 12 months
Time to Treatment failure in subpopulations | Up to 12 months
Tumor response assessed by RECIST or physicians own evaluation | Up to 6 months
  RECIST: Response Evaluation Criteria In Solid Tumors

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan